CLINICAL TRIAL: NCT02908581
Title: Randomized, Open Label Trial of Iron and Folic Acid on Change of Fungal Pattern
Brief Title: Effect of Iron and Folic Acid on Skin Fungal Pattern in Patients With Arsenicosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Prof. Mir Misbahuddin, Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU-010-CT
Record Dates: First submitted 2016-08-28; First posted 2016-09-21 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Chronic Arsenic Poisoning
MeSH Terms: interventions — Iron; Folic Acid; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Active Comparator): 21 Patients Placebo Each tablet by mouth once daily for 12 weeks
  Interventions: Drug: Placebo
- Iron 150 mg and Folic acid 0.5 mg (Experimental): 21 Patients Iron 150 mg and Folic acid 0.5 mg Each tablet by mouth once daily for 12 weeks
  Interventions: Drug: Iron 150 mg and Folic acid 0.5 mg

INTERVENTIONS:
Drug: Placebo — Administered orally once daily
  Other Names: Tablet placebo
  Arms: Placebo
Drug: Iron 150 mg and Folic acid 0.5 mg — Iron will be administered with folic acid orally
  Other Names: Tab Ferrous sulfate and Tablet Folic acid
  Arms: Iron 150 mg and Folic acid 0.5 mg

SUMMARY:
This study will be conducted to observe any change in fungal pattern on skin of arsenicosis patients before and after administration of iron (150 mg) and folic acid (0.5 mg) tablets.

DETAILED DESCRIPTION:
Arsenicosis is remaining as a precarious issue in Bangladesh for the last few decades. The fact of resentment is that this perilous condition still remains unresolved worldwide. So, it has become the demand of era to address this issue. Different diseases are manifested in different way. In arsenicosis melanosis and keratosis are the most common manifestations. The actual mechanism of development of keratosis is unclear. Chronic ingestion of arsenic contaminated water causes accumulation of arsenic in keratin rich tissues like skin, hair, nail and producing characteristic skin manifestations like melanosis and keratosis. Metabolism of arsenic depends on folate pathway and dietary deficiency of folic acid reduced the total arsenic excretion and leads to development of cancer. In different study results shown that folic acid reduces the blood arsenic level. As arsenicosis is a chronic disease condition, fungal infection is more common to them. Moreover the skin fungal pattern in arsenicosis yet not known. Therefore, this study will be conducted to determine is there any change in skin fungal pattern in patients with palmar arsenical keratosis before and after administration of iron and folic acid. Forty two patients with palmar arsenical keratosis will be recruited on the basis of inclusion and exclusion criteria. Twenty one patients will be furnished tablet placebo once daily for 12 weeks without any interruption. Another twenty one patients will be furnished iron (150 mg) and folic acid (0.5 mg) once daily for 12 weeks without any interruption. Water and nail samples will be collected for confirming the diagnosis. Skin sample will be collected two times (before and after giving iron and folic acid) for qualitative analysis of fungi. So, this study will determine any change in fungal pattern after administrating tablet iron and folic acid.

ELIGIBILITY:
Inclusion Criteria: (Patients)

* History of drinking arsenic contaminated water(>50 μg/L) for more than 6 months
* Patients having moderate palmar keratosis
* Patients those voluntarily agree to participate

Exclusion Criteria:

* Pregnant and lactating mother
* Any other chronic diseases like tuberculosis, diabetes mellitus, asthma
* Patient under treatment of arsenicosis on Criteria:

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Changes in the type of fungus in skin surface | [0 weeks (baseline), 12 weeks (end)] [Safety Issue: No]
  Skin swab from five areas of skin (palm, dorsum of the hands, front, back of the chest and axilla) will be taken to see the changes in the type of fungus in skin surface in 12 weeks

SECONDARY OUTCOMES:
Scoring palmar arsenical keratosis | [0 weeks (baseline), 12 weeks (end)] [Safety Issue: No]
  Palmar arsenical keratosis will be scored at 0 week and 12 weeks. The change in the score after 12 weeks following supplementation with folic acid will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Mir Misbahuddin, PhD, Study Director — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh; Priyanka Moitra, MBBS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Laksham Upazilla Health Complex, Comilla, Bangladesh

IPD SHARING:
Plan to Share IPD: No